CLINICAL TRIAL: NCT02918747
Title: P-Gemoxd Regimen Followed by Radiotherapy Versus P-CHOP Regimen Followed by Radiotherapy in ENKTL With Early Stage: a Randomized, Multicenter, Open-label, Phase 2 Study
Brief Title: PEG-ASP+Gemoxd vs. PEG-ASP+CHOP as First-line Chemotherapy to Treatment NK/T-cell Lymphoma With Early Stage
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HNCH-NKT-2016
Record Dates: First submitted 2016-09-25; First posted 2016-09-29 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — pegaspargase; Gemcitabine; Oxaliplatin; Dexamethasone; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- P-Gemoxd (Experimental): Pegaspargase+Gemcitabine+Oxaliplatin+Dexamethasone (PEG-ASP+Gemoxd): Patients received the P-Gemoxd chemotherapy regimen every 3 weeks.
  Pegaspargase 2000U/m2 im day 1, Gemcitabine 800mg/m2 ivdrip 30min day 1 and day 5, Oxaliplatin 85mg/m2 ivdrip day 1, Dexamethasone 15 mg ivdrip, QD, day 1 to day 5.
  IMRT：IMRT is delivered using 6-8 MeV linear accelerator using intensity-modulated radiation treatment planning. The radiation dose is 50 -56grays (Gy) in 25-28 fractions.
  Interventions: Drug: pegaspargase; Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Dexamethasone; Radiation: IMRT
- P-CHOP (Active Comparator): Pegaspargase+Cyclophosphamide+Doxorubicin+Vincristine +Prednisone (P-CHOP)：Patients received the P-CHOP chemotherapy regimen every 3 weeks. Cyclophosphamide 750 mg/m2，ivdrip day 1； doxorubicin 50mg/m 2，ivdrip day 1；vincristine 1.4 mg/m 2(≤2mg），ivdrip day 1; Pegaspargase 2000U/m2 im，day 2 and prednisone (60 mg/m 2 /day) on days 1 to 5 orally.
  IMRT is delivered using 6-8 MeV linear accelerator using intensity-modulated radiation treatment planning. The radiation dose is 50-56 grays (Gy) in 25-28 fractions.
  Interventions: Drug: pegaspargase; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Radiation: IMRT

INTERVENTIONS:
Drug: pegaspargase — P-Gemoxd Arm: 2000U/m2 im on day 1 of each 21 day cycle. Number of Cycles: four.
  P-CHOP Arm: 2000U/m2 im on day 2 of each 21 day cycle. Number of Cycles: four.
  Other Names: Oncaspar
Drug: Gemcitabine — 800mg/m2, ivd on day 1 and 5 of each 21 day cycle. Number of Cycles: four.
  Other Names: Gemzar
  Arms: P-Gemoxd
Drug: Oxaliplatin — 85 mg/m2 ivd on day 1 of each 21 day cycle. Number of Cycles: four
  Other Names: Eloxatin
  Arms: P-Gemoxd
Drug: Dexamethasone — 15 mg, Ivd on day 1 to day 5 of each 21 day cycle. Number of Cycles: four.
  Arms: P-Gemoxd
Drug: Cyclophosphamide — 750 mg/m2，ivdrip day 1 of each 21 day cycle. Number of Cycles: four.
  Arms: P-CHOP
Drug: Doxorubicin — 50mg/m 2，ivdrip day 1 of each 21 day cycle. Number of Cycles: four.
  Arms: P-CHOP
Drug: Vincristine — 1.4 mg/m 2(≤2mg），ivdrip day 1 of each 21 day cycle. Number of Cycles: four.
  Arms: P-CHOP
Drug: Prednisone — 60 mg/m 2 /day orally on days1- 5 of each 21 day cycle. Number of Cycles: four.
  Arms: P-CHOP
Radiation: IMRT — After chemotherapy, if the patients get CR, PR or SD, IMRT is delivered using 6-8 MeV linear accelerator using intensity-modulated radiation treatment planning. The radiation dose is 50 -56grays (Gy) in 25-28 fractions.
  Other Names: intensity-modulated radiation treatment

SUMMARY:
Extranodal natural killer/T-cell lymphoma (ENKTL) is an aggressive subtype of non-Hodgkin's lymphoma and shows extremely poor survival. Several retrospective studies and singe-arm prospective phase 2 studies have shown that pegaspargase combined Gemox or CHOP regimen achieved a promising efficacy in treatment of ENKTL. However, there is no prospective study to compare the efficacy of these two regimens. This prospective pilot study to compare the efficacy and safety of the P-Gemoxd chemotherapy regimen with those of the P-CHOP regimen for stage IE to IIE ENKTL.

DETAILED DESCRIPTION:
Treatment PA-Gemoxd dosages were as follows: days 1 and 5, 30-min intravenous infusion of 800 mg/m2 gemcitabine; day 1, 2-h intravenous infusion of 85 mg/m2 oxaliplatin; day 1, deep intramuscular injection of 2000 U/m2 PEG-ASP at four different sites; d1-5, intravenous infusion of 15mg dexamethasone. The regimen was repeated every 3 weeks for four cycles followed by involved-field radiotherapy after got CR, PR or SD. Three-dimensional conformal radiotherapy was done by linear accelerator at 2.0 grays (Gy) per daily fraction with 5-6 weeks. The involved- field radiation (IFRT) dose was 50-56 Gy.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically confirmed, previously untreated ENKTL with stage I/II (for stage I, the patients should have one of the following risk factors: EBV-DNA > upper limit of normal, lesions beyond nasal, fever, LDH elevation);
2. age range from 18 to 70 years;
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
4. at least one measurable lesion;
5. adequate haematologic function (haemoglobin > 8.0 g/l, absolute neutrophil count > 1500/ml, platelets > 75,000/l),
6. adequate hepatic function (total serum bilirubin ≤ 1.5 times the upper limit of normal, alanine aminotransferase and aspartate aminotransferase ≤ 2.5 times the upper limit of normal),
7. Hepatitis B virus carriers should have normal HBV-DNA copies and should use antiviral drugs. For patients with elevated HBV-DNA, should use antiviral drugs until the HBV-DNA decrease to < the upper limit of normal.
8. adequate renal function (serum creatinine ≤ 1.5 mg/dl, creatinine clearance ≥ 50 ml/min);
9. normal coagulation function and electrocardiogram results.
10. Prior chemotherapy and radiotherapy should have been completed >4 weeks earlier,
11. willingness to provide written informed consent.

Exclusion Criteria:

1. mismatch the inclusion criteria
2. systematic central nervous system involvement, previous or concomitant malignancies and any coexisting medical problems that could cause poor compliance with the study protocol.
3. primary lesion not from the upper respiratory

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-09; Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate（complete remission rate + partial remission rate） | every 6 weeks,up to completion of treatment (approximately 6 months)
  The criteria for the efficacy evaluation (overall response rate and complete remission) of the regimen is according to the following article: Cheson BD, Fisher RI, Barrington SF, et al. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68.
progression free survival | up to end of follow-up-phase (approximately 3 years)
  time from the date of enrollment to date of disease progression, or death of any cause, or date of lost follow-up, whichever comes first
overall survival | up to end of follow-up-phase (approximately 3 years)
  overall survival (OS): time from the date of enrollment to date of death from any cause, or date of lost follow-up, whichever comes first

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events according to Common Terminology Criteria for Adverse Events v3.0 | every 3 weeks,up to completion of treatment (approximately 6 months)
  including hematological safety and non-hematological safety. All the adverse events will be classified according to Common Terminology Criteria for Adverse Events v3.0 (CTCAE)

OTHER OUTCOMES:
Serum Epstein-Barr virus (EBV) DNA copies | every 3 weeks,up to completion of treatment (approximately 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhou, MD., Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No